CLINICAL TRIAL: NCT05868759
Title: Assessment of Preoperative and Postoperative Ankle Kinematics
Acronym: TAR-RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Massimiliano Mosca, Principal Investigator, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TAR-RSA/2020/Sper/IOR
Record Dates: First submitted 2022-05-26; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-05

CONDITIONS: Ankle Osteoarthritis
Keywords: ankle ostearthritis; ankle prosthesis; Roentgen Stereophotogrammetric Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): Candidates for an ankle prosthesis
  Interventions: Radiation: Roentgen Stereophotogrammetric Analysis (RSA); Device: Delos Postural Proprioceptive System (computerized oscillating platform); Diagnostic Test: Modified Star Excursional Balance Tests; Device: Inertial sensors Xsens MVN; Other: American Orthopaedic Foot and Ankle Score (AOFAs); Other: Visual Analogue Scale (VAS); Other: 12-Item Short Form Survey (SF-12)

INTERVENTIONS:
Radiation: Roentgen Stereophotogrammetric Analysis (RSA) — Roentgenstereophotogrammetric analysis (RSA) is a radiographic technique, highly accurate both to evaluate the primary stability of the implant, then the micromovements between bone and implant prosthetic, both for the evaluation of the kinematics of the prosthetic components. The RSA technique in dynamics is able to obtain, with patient in motion, a series of radiographic frames in sequence in two projections, which are captured simultaneously. Each pair of orthogonal projections corresponds to a specific moment of the movement carried out by the patient and will be used to obtain, through dedicated software, a reconstruction three-dimensional instant defined "RSA scenes".
Device: Delos Postural Proprioceptive System (computerized oscillating platform) — The Delos Postural Proprioceptive System uses electronic tilting tables (on a single axis or three axes) with high frequency that allows very short stop and reversal times that allow both to study the proprioception and the patient's response to the modification of movement of the inclined plane
Diagnostic Test: Modified Star Excursional Balance Tests — The Star Excursional Balance Test (SEBT) is a clinical test designed for the evaluation of dynamic physical performance of the tibiotarsica. The first literary references date back to 1998 and the test, remaining in balance with the ankle in the studio, the achievement of the maximum possible distance with the contralateral foot along well-defined axes.
Device: Inertial sensors Xsens MVN — The inertial motion acquisition system Xsens MVN is easy to use and economic to detect the movement of different anatomical districts. MVN is based on inertial sensors in miniature through communication solutions combined with advanced fusion algorithms sensors, using hypotheses of biomechanical models.
  This MVN system is a system of inertial kinematic measurement of the whole body, which incorporates synchronized data. Instant graphic output is provided, including angles of motion articular.
Other: American Orthopaedic Foot and Ankle Score (AOFAs) — American Orthopaedic Foot and Ankle Score (AOFAs) is a clinical trial commonly used in scientific literature which serves to assess, in terms of value from 0 to 100, the autonomy, pain, stability, ankle alignment and back foot of the patient.
Other: Visual Analogue Scale (VAS) — The Visual Analogue Scale (VAS) is a visual representation of the extent of pain that the patient subjectively warns. The VAS is represented by a 10 cm long line in the original version validated, with or without notches at each centimeter. One end indicates the absence of pain and corresponds to 0, the other end indicates the worst pain imaginable and corresponds to 10.
Other: 12-Item Short Form Survey (SF-12) — The 12-Item Short Form Survey (SF-12) is a self-reported outcome measure assessing the impact of health on an individual's everyday life.

SUMMARY:
The objective is to study the joint kinematics of the prosthetic implant, in terms of translation, rotation, Range of motion and proprioception, in patients treated for prosthetic replacement of the ankle, quantitatively and under physiological load conditions.

DETAILED DESCRIPTION:
Patients will be subjected to the same tests at zero time and 9 months after the implantation of the prosthesis, except for RSA which will be performed only 9 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for ankle prosthesis
* Potential party able to provide informed consent and sign the approved Informed Consent Form;
* Male or female patients aged 40 to 80;
* Patients available to perform post-operative rehabilitation according to standard protocol, follow-up visits and radiological investigations scheduled for follow-up up up up to 24 months. In addition, patients who are available to perform all study tests, preoperators and follow-up.

Exclusion Criteria:

* Previous total prosthetic replacement of the ankle (revision surgery);
* Severe pre-operative deformity in valgus or varus (>10 sanguine); BMI>40 kg/m2;
* Pre-existing abnormalities of walking kinematics (amputations, neuro-muscular diseases, polio, hip dysplasia);
* Severe arthrosis of the knee (Kellgren-Lawrence>3);
* Severa coxartrosi (Kellgren-Lawrence>3);
* Previous hip and/or knee prosthesis surgery;
* Total avascular astragalus necrosis or other severe bone loss of the ankle that makes the implantation of standard prosthetic components contraindicated;
* Pregnancy confirmed by positive hcg serum or in vitro diagnostic test or ongoing breastfeeding;
* Active or latent infection of the affected ankle joint or any other systemic infection being treated;
* History of alcoholism, drug or substance abuse intravenously, psychosis, personality disorder/s, poor motivation, emotional or intellectual problems that could make the potential subject unstable for participation in the trial, or any combination of variables which in the opinion of the Principal Investigator should exclude the potential subject;
* Clinically documented acute or chronic pathology, other than the indication for the treatment adopted in this Trial, which could affect life expectancy or make it difficult to interpret the outcome of the potential subject in accordance with the Protocol (e.g., renal, hepatic, cardiac, endocrine, haematological, autoimmune, bone metabolism, crystal deposits or neoplasms);
* Potential subjects with medical conditions that interfere with the ability to participate in a standardized rehabilitation program;
* Participation in any other trial of another drug or experimental device within 60 days prior to the screening visit or administration of that drug or device during the course of this trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Roentgenstereophotogrammetric analysis | 9 months
  Roentgenstereophotogrammetric analysis (RSA) is a radiographic technique, highly accurate both to assess the primary stability of the implant, and therefore the micromovements between bone and prosthetic implant, and for the evaluation of the kinematics of the prosthetic components.
  Using reference points it is possible to measure the micro-movements that occur between several contiguous elements

SECONDARY OUTCOMES:
evaluation of range of motion (degree) | at baseline (Day0)
  motion tracker
evaluation of range of motion (degree) | 9 months
  motion tracker
Delos Postural Proprioceptive System | at baseline (Day0)
  The patients will be analyzed pre and postoperatively using a computerized oscillating platform that shows the response of the foot as an adaptation to the ground. The result is expressed through stability index (%) compared to the average of the population
Delos Postural Proprioceptive System | 9 months
  The patients will be analyzed pre and postoperatively using a computerized oscillating platform that shows the response of the foot as an adaptation to the ground. The result is expressed through stability index (%) compared to the average of the population
modified Star Excursional Balance Test (mSEBT) functional test | at baseline (day 0)
  mSEBT: best value resulting from the 3 equilibrium tests standardized for the length of the limb. The tests consist in reaching the greater distance with a foot along three (inverted Y-shaped) axes with between them an angle of 90 ° (rear) and two of 135 ° (antero-medial and anterior-lateral) while the opposite foot remains still on the ground
modified Star Excursional Balance Test (mSEBT) functional test | 9 months
  mSEBT: best value resulting from the 3 equilibrium tests standardized for the length of the limb. The tests consist in reaching the greater distance with a foot along three (inverted Y-shaped) axes with between them an angle of 90 ° (rear) and two of 135 ° (antero-medial and anterior-lateral) while the opposite foot remains still on the ground
American Orthopaedic Foot & Ankle score (AOFAs) questionnaire | at baseline (Day0)
  AOFAs: values from 0 to 100 dependent on limitations in performing activities
American Orthopaedic Foot & Ankle score (AOFAs) questionnaire | 9 months
  AOFAs: values from 0 to 100 dependent on limitations in performing activities
Short Form Health Survey - 12 questionnaire | at baseline (Day0)
  SF12: personal assessment of one's state of health using multiple-answer questions with different values for each question.
Short Form Health Survey - 12 questionnaire | 9 months
  SF12: personal assessment of one's state of health using multiple-answer questions with different values for each question.

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Riva D, Bianchi R, Rocca F, Mamo C. Proprioceptive Training and Injury Prevention in a Professional Men's Basketball Team: A Six-Year Prospective Study. J Strength Cond Res. 2016 Feb;30(2):461-75. doi: 10.1519/JSC.0000000000001097. PMID 26203850
- [Result] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Result] Gougoulias NE, Khanna A, Maffulli N. History and evolution in total ankle arthroplasty. Br Med Bull. 2009;89:111-51. doi: 10.1093/bmb/ldn039. Epub 2008 Nov 13. PMID 19008282
- [Result] Selvik G. Roentgen stereophotogrammetry. A method for the study of the kinematics of the skeletal system. Acta Orthop Scand Suppl. 1989;232:1-51. PMID 2686344